CLINICAL TRIAL: NCT05393336
Title: Comparison of V-sitting Posture Stabilization and Modified Clamshell Exercises on Pain and Disability in Patients With Non-specific Chronic Low Back Pain.
Brief Title: V-sitting Posture Stabilization Versus Modified Clamshell in Patients With Non-specific Chronic Low Back Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0104
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Non-specific Chronic Low Back Pain
Keywords: low back pain; disability; pain intensity; chronic pain
MeSH Terms: conditions — Low Back Pain; Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- V-sitting posture stabilization (Experimental): V sitting exercises will be administered where patients will be asked to lift the torso and legs while engaging the core and abdominal muscles.
  Interventions: Other: V-sitting posture stabilization
- modified clamshell exercises (Experimental): Participants will perform modified clamshell exercises monitored visually and using a stabilizer pressure biofeedback unit.
  Interventions: Other: Modified clamshell exercises

INTERVENTIONS:
Other: V-sitting posture stabilization — 15 patients will be given a hot pack with TENS for 15 minutes. Followed by static stretching of the gluteus, hamstrings, and Iliopsoas muscles for 10 to 30 seconds hold and 2 to 4 repetitions. Then the patient will perform the V-sitting exercise for 10 seconds starting with 5 repetitions and progressing to 15 overtime. Each patient will receive treatment for 6 days per week and 6 weeks.
  Arms: V-sitting posture stabilization
Other: Modified clamshell exercises — 15 patients will be given a hot pack with TENS for 15 minutes. Followed by static stretching of the gluteus, hamstrings, and Iliopsoas muscles for 10 to 30 seconds hold and 2 to 4 repetitions. Then the patient will perform the modified clamshell exercise for 10 seconds starting with 5 repetitions and progressing to 15 overtime. Each patient will receive treatment for 6 days per week and 6 weeks.
  Arms: modified clamshell exercises

SUMMARY:
The aim of this study is to compare the v-siting posture stabilization and clamshell exercises on pain and disability in patients with non-specific chronic low back pain.

DETAILED DESCRIPTION:
Chronic low back pain (LBP) is a common musculoskeletal pain disorder that affects most adults and has the highest prevalence among other chronic musculoskeletal pain disorders. Non-traumatic lower back pain can have different etiologies: intervertebral disc related, vertebral body related, and facet joint related and sacroiliac joint related. Non-specific low back pain affects people of all ages and is a leading contributor to disease burden worldwide. Non-specific low back pain does not have a known pathoanatomical cause. Treatment of non-specific chronic low back pain includes manual therapy, exercise therapy, massage, acupuncture, yoga, cognitive behavioral therapy, and intensive interdisciplinary treatment.

Previous studies have compared the effects of different exercise therapies, other treatment modalities, osteopathic techniques, manual therapies, and yoga and eurhythmy therapy for the management of low back pain. There is very little literature found to evaluate the effects of single movement technique V-sitting exercises and modified clamshell exercises in the management of non-specific chronic low back pain. Previous literature showed less treatment sessions and follow up periods as they are barrier to see the exact picture of effects of treatment protocol followed. In contrast longer duration of treatment regime allow deep insight of the effects of the main treatment body. This study will fulfill these literature gaps. This study will find the comparative effects of V-sitting posture stabilization and Modified Clamshell exercises in the treatment of non-specific chronic low back pain with more treatment sessions in both genders.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-specific low back pain for more than 3 months
* Subjects being able to sustain 5 seconds of isometric hip abduction in the side-lying position
* Negative Crossed Straight leg raise test
* Negative Straight leg raise test

Exclusion Criteria:

* Metabolic Bone disease (Osteoporosis)
* Any History of Hip pathology
* History of trauma
* History of systemic disease (Rheumatologic disorders, spondylitis, spinal cord disease)
* Radiculopathy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
NPRS for pain | 6th week
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
RMQ for pain and disability | 6th week
  The Roland-Morris Questionnaire (RMQ) is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale. For example, at the beginning of treatment, a patient's score was 12 and, at the conclusion of treatment, their score was 2 (10 points of improvement), we would calculate an 83% (10/12 x 100) improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman Bashir, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwok BC, Lim JXL, Kong PW. The Theoretical Framework of the Clinical Pilates Exercise Method in Managing Non-Specific Chronic Low Back Pain: A Narrative Review. Biology (Basel). 2021 Oct 25;10(11):1096. doi: 10.3390/biology10111096. PMID 34827088
- [Background] Cho JH, Lee KH, Lim ST. Aged Lumbar Extension Strength of Chronic Low Back Pain in Korean Population of 10-80 Years. Iran J Public Health. 2020 Oct;49(10):1894-1901. doi: 10.18502/ijph.v49i10.4692. PMID 33346210
- [Background] Popescu A, Lee H. Neck Pain and Lower Back Pain. Med Clin North Am. 2020 Mar;104(2):279-292. doi: 10.1016/j.mcna.2019.11.003. Epub 2019 Dec 20. PMID 32035569
- [Background] Clark JR, Nijs J, Smart K, Holmes P, Yeowell G, Goodwin PC. Prevalence of Extreme Trait Sensory Profiles and Personality Types in Nonspecific Chronic Low Back Pain with Predominant Central Sensitization: Secondary Analysis of an International Observational Study. Pain Physician. 2019 May;22(3):E181-E190. PMID 31151341
- [Background] Tanabe H, Akai M, Doi T, Arai S, Fujino K, Hayashi K; for Low back-pain Traction Therapy (LTT) Study. Immediate effect of mechanical lumbar traction in patients with chronic low back pain: A crossover, repeated measures, randomized controlled trial. J Orthop Sci. 2021 Nov;26(6):953-961. doi: 10.1016/j.jos.2020.09.018. Epub 2021 Mar 27. PMID 33785233
- [Background] van Dillen LR, Lanier VM, Steger-May K, Wallendorf M, Norton BJ, Civello JM, Czuppon SL, Francois SJ, Roles K, Lang CE. Effect of Motor Skill Training in Functional Activities vs Strength and Flexibility Exercise on Function in People With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Neurol. 2021 Apr 1;78(4):385-395. doi: 10.1001/jamaneurol.2020.4821. PMID 33369625
- [Background] Krause F, Niederer D, Banzer W, Vogt L. Medical exercise and physiotherapy modes and frequency as predictors for a recurrence of chronic non-specific low back pain. J Back Musculoskelet Rehabil. 2021;34(4):665-670. doi: 10.3233/BMR-200149. PMID 33749637
- [Background] Dal Farra F, Risio RG, Vismara L, Bergna A. Effectiveness of osteopathic interventions in chronic non-specific low back pain: A systematic review and meta-analysis. Complement Ther Med. 2021 Jan;56:102616. doi: 10.1016/j.ctim.2020.102616. Epub 2020 Nov 13. PMID 33197571
- [Background] Sanchis-Sanchez E, Lluch-Girbes E, Guillart-Castells P, Georgieva S, Garcia-Molina P, Blasco JM. Effectiveness of mechanical diagnosis and therapy in patients with non-specific chronic low back pain: a literature review with meta-analysis. Braz J Phys Ther. 2021 Mar-Apr;25(2):117-134. doi: 10.1016/j.bjpt.2020.07.007. Epub 2020 Aug 4. PMID 32773288